CLINICAL TRIAL: NCT06207435
Title: Community Support Program for Lung Cancer Screening
Acronym: LCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UPCC 07523; 852598 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2023-12-20; First posted 2024-01-17 (Actual); Results first posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer; Behavior
Keywords: screening adherence
MeSH Terms: conditions — Lung Neoplasms; Behavior | interventions — Transportation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- West Philadelphia Residents (Experimental): For eligible residents of West Philadelphia, patients are contacted by Community Support Program Representative and offered free Lyft transportation to and from appointment. If patient has other questions about their upcoming appointment (location, time, etc.), Patient Navigator assists in answering questions
  Interventions: Behavioral: Transportation
- Non West Philadelphia Residents (No Intervention): For patients outside West Philadelphia, no contact is made and no free transportation is provided. Research coordinator logs their appointment attendance after the appointment date in question.

INTERVENTIONS:
Behavioral: Transportation — Eligible patients are contacted and offered free transportation to and from their upcoming appointment.
  Arms: West Philadelphia Residents

SUMMARY:
The research study aims to create a program for lung cancer screening attendance

DETAILED DESCRIPTION:
The overall objective of this project is to demonstrate the impact of a community support program (CSP) on improving adherence to LCS follow-up guidelines in an urban environment. The project aims to collaborate with community partners to develop an infrastructure and iterative process to provide social support to community members that facilitates obtaining their follow-up LDCT for LCS. It utilizes novel population level data that includes geospatial analysis of neighborhood-level data of patients residing in Philadelphia who have received a LDCT for LCS. This allows for targeted community level interventions and the ability to evaluate impact on a population level.

A Community Support Program Representative will reach out to eligible patients via telephone. The CSP Representative and Patient Navigator will communicate with consented patient directly, assist with travel and the appointment. The PN will log the date of the appointment, zip code of the patient and the adherence (or lack of) of the appointment completion. We will utilize Lyft transportation vouchers to provide rides to participants from their home location in West Philadelphia to and from the Penn Medicine downtown hospital locations on the day of their LDCT.

ELIGIBILITY:
Inclusion Criteria:

* Upcoming or missed follow-up LDCT (low dose CT)
* West Philadelphia resident
* Between 18-89 years' old

Exclusion Criteria:

* No upcoming LDCT
* Lives outside West Philadelphia
* Outside age range

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farouk Dako, MD, MPH, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- West Philadelphia CSP Participants: For eligible residents of West Philadelphia, patients are contacted by Community Support Program Representative and offered free Lyft transportation to and from appointment. If patient has other questions about their upcoming appointment (location, time, etc.), Patient Navigator assists in answering questions. This group opted into the CSP.
- West Philadelphia Non CSP Participants: For eligible residents of West Philadelphia, patients are contacted by Community Support Program Representative and offered free Lyft transportation to and from appointment. If patient has other questions about their upcoming appointment (location, time, etc.), Patient Navigator assists in answering questions. This group did not opt into the CSP.
- Southwest Philadelphia Residents: For patients outside West Philadelphia, no contact is made and no free transportation is provided. Research coordinator logs their appointment attendance after the appointment date in question.
Period: Overall Study
Arm/Group | West Philadelphia CSP Participants | West Philadelphia Non CSP Participants | Southwest Philadelphia Residents
Started | 26 | 165 | 51
Completed | 26 | 165 | 51
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | West Philadelphia CSP Participants | West Philadelphia Non CSP Participants | Southwest Philadelphia Residents | Total
Number analyzed (Participants) | 26 | 165 | 51 | 242
Age, Customized [Number; unit: participants]
  Age 18-89 | 26 | 165 | 51 | 242
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 98 | 28 | 144
  Male | 8 | 67 | 23 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 26 | 162 | 51 | 239
  Unknown or Not Reported | 0 | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 2
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 26 | 149 | 48 | 223
  White | 0 | 11 | 3 | 14
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 26 | 165 | 51 | 242
Scheduled Lung Cancer Screening [Number; unit: participants] | 26 | 165 | 51 | 242

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Scheduled Lung Cancer Screening Appointments Attended by Participants
Description: The Primary Outcome measures the rate of appointment attendance across three groups: West Philadelphia CSP Participants (eligible West Philadelphia residents who opted into the CSP), West Philadelphia Non CSP Participants (eligible West Philadelphia residents who did not opt into the CSP), and Southwest Philadelphia Residents (patients who did not receive an option to participate in the CSP).
Time Frame: 12 months
Measure: Number; unit: % of lcs appointment attendance
Groups:
- West Philadelphia CSP Participants: West Philadelphia CSP Participants For eligible residents of West Philadelphia, patients are contacted by Community Support Program Representative and offered free Lyft transportation to and from appointment. If patient has other questions about their upcoming appointment (location, time, etc.), Patient Navigator assists in answering questions. This group opted into the CSP.
Arm/Group | West Philadelphia CSP Participants | West Philadelphia Non CSP Participants | Southwest Philadelphia Residents
Number analyzed (Participants) | 26 | 165 | 51
% of lcs appointment attendance | 88 | 68 | 64

2. Secondary Outcome: Percentage of CSP Enrollment
Description: The Secondary outcome is a measurement of the percentage of eligible participants (West Philadelphia residents) who chose to opt into the CSP (as opposed to eligible participants who did not).
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | West Philadelphia Residents
Number analyzed (Participants) | 191
percentage of participants | 14

ADVERSE EVENTS:
Description: Adverse events were not assessed. The only intervention provided was optional transportation for a clinical scan already scheduled by the patient's care team.
Arm/Group | West Philadelphia Residents | Non West Philadelphia Residents
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/35/NCT06207435/Prot_SAP_001.pdf
  • Informed Consent Form (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT06207435/ICF_002.pdf